CLINICAL TRIAL: NCT07084636
Title: Comparative Study of Video Laryngeal Mask and Endotracheal Intubation in Airway Management in Patients Undergoing Tympanoplasty Surgery.
Brief Title: Comparative of Video Laryngeal Mask and Endotracheal Intubation in Patients Undergoing Tympanoplasty Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GOKAEK 2024/21/10
Record Dates: First submitted 2025-06-23; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Tympanoplasty Surgery; Laryngeal Mask Airway
Keywords: tympanoplasty; video laryngeal mask; airway; intubation; general anesthesia
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Laryngeal Mask Airway (Active Comparator): In this group, after 3 minutes of preoxygenation, 2 mg/kg propofol will be administered intravenously. A laryngeal mask will be placed after induction, the cuf will be inflated and fixed with a cuf manometer.
  Interventions: Other: Video Laryngeal Mask
- Group Endotracheal Tube (Active Comparator): In this group, after 3 minutes of preoxygenation, 2 mg/kg propofol will be administered intravenously, 1 mcg/kg fentanyl will be administered intravenously. Additionally, 0.6 mg/kg rocuronium will be administered intravenously and endotracheal intubation will be performed, and the cuff will be inflated and fixed with a cuff manometer.
  Interventions: Other: Endotracheal intubation

INTERVENTIONS:
Other: Video Laryngeal Mask — Video laryngeal mask will be used in this group
  Arms: Group Laryngeal Mask Airway
Other: Endotracheal intubation — Endotracheal intubation will be performed in this group.
  Arms: Group Endotracheal Tube

SUMMARY:
The effects of video laryngeal mask and endotracheal intubation on hemodynamic parameters and the development of postoperative respiratory complications in participants scheduled for tympanoplasty will be evaluated.

DETAILED DESCRIPTION:
Procedures to be performed under general anesthesia are performed by placing endotracheal intubation and laryngeal mask in the airway. Video Laryngeal Mask (LMA) combines the upper glottic airway device with video laryngoscope tracheal intubation. LMA placement and tracheal intubation can be visualized, LMA position can be continuously monitored during the operation, and adverse events such as LMA displacement can be managed in a timely manner. Studies have shown that video LMA has extraordinary advantages in airway management. This study aimed to compare video LMA and endotracheal intubation in participants who will undergo tympanoplasty surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-75
* Participants with ASA I-II-III
* Cases with surgery duration of less than two hours

Exclusion Criteria:

* Participants under 18 years of age
* Participants who are pregnant
* Participants with a difficult airway diagnosis
* Participants with a mouth opening of less than 4 cm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-17 (Actual)

PRIMARY OUTCOMES:
Time to Effective Airway | Baseline
  The time to achieve an effective airway was defined as the time between removing the face mask, attaching the airway device, and obtaining 3 square wave capnograph traces with manual ventilation.

SECONDARY OUTCOMES:
Number of attempts taken for successful placement of airway device | Baseline
  Number of attempts needed for successful placement of either the SaCoVLM™ video laryngeal mask airway the tracheal tube, as assigned
Haemodynamic response to insertion of airway device | Baseline, 1st minute, 5th minute
  Systolic blood pressure and heart rate at 0th minute, 1st minute 5th minute, starting from the time the face mask was removed from the patient's face.
Displacement of the SaCoVLM™ video laryngeal mask in head position | Baseline
  Effect of Head Rotation During Tympanoplasty on laryngeal visibility with the SaCoVLM™ Laryngeal Mask during head rotation
Incidence of post-operative sore throat | 24 hours after surgery
  postoperative sore throat will be recorded at 1st hour, 6th hour, 12th hour, 18th hour, 24th hour

CONTACTS AND LOCATIONS:
Overall Officials: HATİCE SELÇUK KUŞDERCİ, asst prof, Study Director — SAMSUN UNİVERSITY
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Sun Y, Huang L, Xu L, Zhang M, Guo Y, Wang Y. The Application of a SaCoVLMTM Visual Intubation Laryngeal Mask for the Management of Difficult Airways in Morbidly Obese Patients: Case Report. Front Med (Lausanne). 2021 Nov 18;8:763103. doi: 10.3389/fmed.2021.763103. eCollection 2021. PMID 34869469
- [Background] Yan CL, Chen Y, Sun P, Qv ZY, Zuo MZ. Preliminary evaluation of SaCoVLM video laryngeal mask airway in airway management for general anesthesia. BMC Anesthesiol. 2022 Jan 3;22(1):3. doi: 10.1186/s12871-021-01541-0. PMID 34979936
- [Background] Choi WJ, Kim YH. The influence of head rotation on ProSeal laryngeal mask airway sealing during paediatric myringotomy. Anaesth Intensive Care. 2007 Dec;35(6):957-60. doi: 10.1177/0310057X0703500617. PMID 18084990